CLINICAL TRIAL: NCT02771236
Title: Clinical and Molecular Studies in Families With Inherited Eye Disease
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160104; 16-EI-0104
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-06-13

CONDITIONS: Inherited Eye Disease
Keywords: Genetics; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Participants with cataracts: Participants with cataracts
- Participants with corneal dystrophies: Participants with corneal dystrophies
- Participants with glaucoma: Participants with glaucoma or other anterior chamber anomalies
- Participants with lens refractive errors: Participants with lens refractive errors including myopia and hyperopia
- Participants with retinal degenerations: Participants with retinal degenerations

SUMMARY:
Background:

Genes are the basic units of heredity. When genes are changed, certain cells don t work like they should. Researchers want to try to better understand the genetic conditions that are linked with inherited eye diseases.

Objective:

To try to identify the genes linked to the development of inherited eye diseases.

Eligibility:

People ages 4 and older who have or have a family member with an inherited eye disease

Design:

Participants will be screened with medical history and medical records.

Participants will have one visit that will take 3-4 hours. This will include:

Medical and family history

Eye exam: This includes the pupil being dilated.

Electroretinography: A small electrode is taped to the forehead. Participants sit in the

dark with their eyes patched for 30 minutes. Then numbing drops and contact lenses are put in

the eyes. They will watch flashing lights.

Blood tests

Saliva sample: They will spit into a container or have the inside of their cheek swabbed.

Genetic testing will be done on participants blood or saliva.

Participants may meet with the researchers to discuss their genetic tests.

DETAILED DESCRIPTION:
Objective: This project, Clinical and Molecular Studies in Families with Inherited Eye Disease will study inherited eye diseases, both Mendelian and complex age related inherited eye diseases, in families of many nationalities and ethnic backgrounds in order to identify the genes that, when mutated, cause inherited eye diseases and the pathophysiology through which they act. Among the diseases studied will be cataracts, corneal dystrophies and other corneal diseases, retinal degenerations, myopia and other anterior chamber defects, and glaucoma.

Study Population: Families and individuals of many nationalities and ethnic backgrounds. We will study a maximum of 5,000 participants and family members.

Design: The study consists of ascertaining individuals and especially families with multiple individuals, affected by both congenital and age related inherited eye diseases. These participants and their families will undergo detailed ophthalmological examinations to characterize their visual system and determine their affectation status. A blood sample will be collected from each individual for isolation of DNA and in some individuals for lymphoblastoid transformation to establish a renewable source of DNA. Linkage analysis, association analysis, physical mapping, and mutational screening will be carried out to identify the specific gene and the mutations in it that are associated with inherited eye disease in the family. Mutation screening may involve Sanger sequencing if a small number of candidate genes are identified, or whole genome or whole exome sequencing if more genes remain as viable candidates after the initial analysis. If necessary, the gene product will be characterized biochemically. Blood samples may also be used to complete analyses such as: hemoglobin A1c (HbA1c), fasting blood glucose, and glucose tolerance tests. The study will enroll participants at NEI and collaborating institutions.

Outcome Measures: Linkage will be determined using the lod score method, association will be determined using standard statistical procedures to estimate p values, and mutations in specific genes will be assessed using a combination of residue conservation, blosum score, bioinformatic prediction of structural damage to the protein, and molecular modeling. Assessment of biochemical, metabolic, and physiological effects of these mutations will be individualized to the specific case.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable;

1. Participant must be four years of age or older.
2. Participant must understand and sign the protocol s informed consent document.
3. Individuals or family members of individuals with inherited eye diseases, either congenital, childhood, or age related.
4. All participants must be able to cooperate with study examination and phlebotomy.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present:

1. Participant has a disease, infection, or trauma that mimics inherited cataracts, retinal degenerations, glaucoma, etc.
2. Participant has a significant active infection (an infection requiring treatment as determined by the investigator) or a history of chronic or recurrent infections.
3. Participant requires sedation for study purposes.

Ages: 4 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with inherited eye diseases.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-10-04 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Document the clinical and genetic features of Mendelian and age related visual disorders | Study duration
  Provide improved diagnosis and categorization of inherited visual disorders and should eventually suggest rationales for prevention or delay of both Mendelian and complex eye diseases

CONTACTS AND LOCATIONS:
Overall Officials: James F Hejtmancik, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (10):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Duke University Eye Center, Durham, North Carolina
- Eye Research Institute, Zhongshan Ophthalmic Center, Sun Yat Sen University, Guangzhou, China
- Aravind Medical Research Foundation, Madurai, India
- Seconda Universita di Napoli, Napoli, Italy
- National Centre of Excellence in Molecular Biology, University of the Punjab, Lahore, Pakistan
- University of the Philippines, Manila, Philippines
- The Filatov Institute of Eye Disease and Tissue Therapy of the National Academy, Odesa, Ukraine
- University of Exeter, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-EI-0104.html